CLINICAL TRIAL: NCT04608370
Title: Effects of Transcranial Photobiomodulation Intervention on Working Memory and Functional Brain Networks for Healthy Older Adults
Brief Title: Transcranial Photobiomodulation Intervention for Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XuanwuH 2 (Other)
Collaborators: Beijing Normal University (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HanYingsc4
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Transcranial Photobiomodulation; Intervention; Functional Near-infrared Spectroscopy; Working Memory; Healthy Older Adults
Keywords: Intervention; Neuroimaging; Working memory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tPBM session group (Experimental): Participants in the active tPBM group will take active tPBM session, which include 12 minutes active tPBM by a 1064nm laser to the left forehead , 6 minutes resting-state fNIRS measurement, and 8 minutes digital n-back task-an ubiquitous cognitive task for working memory.
  Interventions: Behavioral: Active tPBM session
- Sham tPBM session group (Active Comparator): Participants in the sham tPBM group will take sham tPBM session, which include 12 minutes sham tPBM by a 1064nm laser to the left forehead , 6 minutes resting-state fNIRS measurement, and 8 minutes digital n-back task-an ubiquitous cognitive task for working memory.
  Interventions: Behavioral: Sham tPBM session

INTERVENTIONS:
Behavioral: Active tPBM session — In this project, taking the method of random, double blindness and control, participants in the active tPBM group will take active tPBM session. After that, N-back tests and neuroimaging biomarkers will be compared between active tPBM group and sham tPBM group.
  Arms: Active tPBM session group
Behavioral: Sham tPBM session — In this project, taking the method of random, double blindness and control, participants in the sham tPBM group will take sham tPBM session. After that, N-back tests and neuroimaging biomarkers will be compared between active tPBM group and sham tPBM group.
  Arms: Sham tPBM session group

SUMMARY:
Transcranial photobiomodulation (tPBM) is a novel, non-invasive neurostimulation technique, which has shown compelling potential for cognitive improvement. Increasing neuroimaging studies have demonstrated that functional brain network models would sensitively and comprehensively delineate action mechanisms of multiple neurostimulation techniques. However, the action mechanism of tPBM based on functional brain network remain largely unknown. In this project, the investigators aim to investigate the effectiveness of tPBM on working memory for healthy older adults. Taking the randomized, single-blind controlled method, participants in the active tPBM group will take active tPBM, and those in the sham tPBM group will take sham tPBM. After that, the investigators will investigate the changes of working. Furthermore, based on the neuroimaging technique, the regulatory mechanism of tPBM in intervening older adults will be revealed from the perspective of altered brain functional networks. This study will provide evidence for understanding whether the tPBM has the potentially therapeutic effect on cognitive function for healthy older adults as a non-drug treatment, and further elucidating the potential brain mechanism, which are of great values in solving scientific and clinical practice issues.

DETAILED DESCRIPTION:
An astonishing rise in the prevalence of cognitive decline and dementia in older adults was witnessed in recent years, which renders investigations of cognitive intervention especially urgent and vital. Transcranial photobiomodulation (tPBM) is now considered as a potentially non-pharmacologic intervention for cognitive decline and has attracted the interest of researchers. However, there are few existing studies involving the mechanism of tPBM on brain functional networks.

Sixty healthy older participants will be recruited in this randomized, single-blind controlled trial. Each group had thirty participants.Participants in the active tPBM group will take active tPBM and those in the sham tPBM group will take sham tPBM. After that, the investigators will investigate the changes of working memory, which is the primary outcome. Furthermore, based on the neuroimaging technique of functional near-infrared spectroscopy (fNIRS), the regulatory mechanism of tPBM in intervening older adults will be revealed from the perspective of altered brain functional networks.

This study will provide evidence for understanding whether the tPBM has the potentially therapeutic effect on cognitive function for healthy older adults as a non-drug treatment, and further elucidating the potential brain mechanism, which are of great values in solving scientific and clinical practice issues.

ELIGIBILITY:
Inclusion Criteria:

* 50-79 years old, right-handed and Mandarin-speaking subjects;
* Normal age-adjusted, gender-adjusted and education-adjusted performance on standardised cognitive tests

Exclusion Criteria:

* Current diagnosis with mild cognitive decline or dementia;
* Current major psychiatric diagnoses such as severe depression and anxiety;
* Other neurological conditions (e.g., cerebrovascular disease, brain tumors, Parkinson's disease, encephalitis, or epilepsy)
* Other diseases which could cause cognitive decline (e.g., thyroid dysfunction, severe anemia, syphilis, or HIV)

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Working memory | 24 hours
  N-back task is one of the most classic cognitive to study working memory (Bopp and Verhaeghen, 2020). During this task, participants are asked to decide if a digit appearing on a screen is the same as the digit that appeared n stimuli earlier (n-back). Working memory load varies with n between blocks. In our study, the digit (0 to 9) was randomly presented on a screen for 1 seconds every 2 seconds and a total of 20 digit formed one trial. The whole task consists of three blocks, and each of block includes 3 trials -sequentially 1-back, 2-back, 3-back. The presentation of n-back were generated by E-Prime 3. Mean accuracy and reaction time for correct trials are used as n-back performance indicators.

SECONDARY OUTCOMES:
FNIRS-based brain functional networks changes | 24 hours
  The brain functional activity data will be collected using functional near-infrared spectroscopy (fNIRS) technique. The investigators will compare the changes of brain functional networks based on the measure of oxyhemoglobin concentration signal with relatively high signal to noise ratio (SNR) in two groups, in order to reveal the regulatory mechanism of the tPBM in intervening older persons.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Department of Neurolgy, Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The information of neuropsychological tests will be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: When summary data are published or starting 6 months after publication
Access Criteria: The information of neuropsychological tests data will be shared.